CLINICAL TRIAL: NCT03217591
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of IW-1973 in Patients With Type 2 Diabetes With Albuminuria Treated With Renin-Angiotensin System Inhibitors
Brief Title: A Study to Evaluate the Soluble Guanylate Cyclase (sGC) Stimulator IW-1973 in Diabetic Nephropathy / Diabetic Kidney Disease as Measured by Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Collaborators: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1973-203
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes Mellitus With Diabetic Nephropathy
MeSH Terms: interventions — praliciguat

STUDY DESIGN:
Intervention Model Description: Phase 2, randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IW-1973 Low Dose (Experimental): Administered daily for 12 weeks
  Interventions: Drug: IW-1973
- IW-1973 High Dose (Experimental): Administered daily for 12 weeks
  Interventions: Drug: IW-1973
- Placebo (Placebo Comparator): Placebo to match experimental drug administered daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-1973 — Oral Tablet
  Arms: IW-1973 Low Dose
Drug: IW-1973 — Oral Tablet
  Arms: IW-1973 High Dose
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of IW-1973 in patients with type 2 diabetes mellitus with albuminuria who are on a stable regimen of renin-angiotensin system inhibitors.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is an ambulatory male or female from 25 to 75 years old at the Screening Visit.
* Patient has type 2 diabetes diagnosed by a physician or nurse practitioner ≥6 months before the Screening Visit, has been on ≥1 antihyperglycemic medication for ≥12 weeks preceding the Randomization Visit, and has been on a stable regimen (ie, same drug and same dose) of ≥1 antihyperglycemic medication for ≥28 days preceding the Randomization Visit. (Modification of short-acting insulin throughout the Screening Period will not affect eligibility.)
* Patient has been on a stable regimen (ie, same drug and dose) of antihypertensive medications, which must include an angiotensin-converting enzyme inhibitor (ACEi) or an angiotensin receptor blocker (ARB), for ≥28 days preceding the Randomization Visit and is expected to remain on their regimen through the Follow-up Visit.
* Patient has the following:

  1. Estimated glomerular filtration rate (eGFR) 30 to 75 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation (1) at the Screening and Baseline Visits
  2. Urine albumin-to-creatinine ratio (UACR) >200 mg/g at the Screening and Baseline Visits and <5000 mg/g at Screening and Baseline Visits
  3. Serum albumin >3.0 g/dL at the Screening and Baseline Visits
  4. Hemoglobin A1c (HbA1c) ≤11% at the Screening and Baseline Visits
  5. Systolic blood pressure (BP) of 110 to 160 mm Hg at the Screening and Baseline Visits
* Women of childbearing potential must have a negative pregnancy test prior to randomization and must agree to use protocol-specified contraception from the Screening Visit through 60 days after the final dose of study drug.
* Male patients must be surgically sterile by vasectomy (conducted ≥60 days before the Screening Visit or confirmed via sperm analysis) or must agree to use protocol-specified contraception from the Screening Visit through 60 days after the final dose of study drug.
* Other inclusion criteria per protocol.

Key Exclusion Criteria:

* Patient has a history of secondary hypertension (ie, renal artery stenosis, primary aldosteronism, or pheochromocytoma).
* Patient has a body mass index (BMI) <20 or >45 kg/m2 at the Screening Visit.
* Patient has a history of platelet dysfunction, hemophilia, von Willebrand disease, coagulation disorder, other bleeding diathesis, or significant, nontraumatic bleeding episode(s), such as from a gastrointestinal source.
* Patient has hepatic impairment defined as Child-Pugh A, B, C.
* Patient has significant comorbidities (eg, malignancy, advanced liver disease, pulmonary hypertension, pulmonary fibrosis, lung disease requiring supplemental oxygen) or other significant conditions that, in the Investigator's opinion, would limit the patient's ability to complete or participate in this clinical study; has been hospitalized for cardiovascular, renal, or metabolic cause in the 3 months before the Screening Visit; or has a life expectancy of less than 1 year.
* Patient has had prior dialysis, renal transplant, or planned renal transplant.
* Patient has clinically active, symptomatic, or unstable coronary artery or heart disease within the 3 months before the Screening Visit, defined as 1 of the following:

  1. Hospitalization for myocardial infarction (MI), unstable angina, or heart failure
  2. New-onset angina with positive functional study or coronary angiogram revealing stenosis
  3. Coronary revascularization procedure
* Patient has a history of clinically significant hypersensitivity or allergies to any of the inactive ingredients contained in the active or placebo drug products.
* Patient has previously received IW-1973 in a study, or received an investigational drug during the 30 days or 5 half-lives of that investigational drug (whichever is longer) before the Screening Visit, or is planning to receive another investigational drug at any time during the study.
* Patient is taking specific inhibitors of phosphodiesterase 5 (PDE5), nonspecific inhibitors of PDE5 (including dipyridamole and theophylline), any supplements for the treatment of erectile dysfunction, riociguat, or nitrates or nitric oxide (NO) donors in any form. These medications and supplements are prohibited from 7 days before Randomization through the duration of the study.
* Patient is taking strong cytochrome P450 3A (CYP3A) inhibitors (eg, ketoconazole, indinavir, nelfinavir, ritonavir, saquinavir, clarithromycin, telithromycin, itraconazole, and nefazodone). These medications are prohibited 14 days before Randomization through the duration of the trial.
* Other exclusion criteria per protocol.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, MD MPH, Study Director — Cyclerion Therapeutics, Inc.
Locations (54):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Institute of Renal Research, Chula Vista, California
  - St. Joseph Heritage Healthcare (St. Jude Hospital DBA), Fullerton, California
  - California Institute of Renal Research, La Mesa, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - American Institute of Research, Los Angeles, California
  - Academic Medical Research Institute, Los Angeles, California
  - California Medical Research Associates, Inc. (CMRA), Northridge, California
  - Riverside Nephrology Physicians, Inc., Riverside, California
  - California Kidney Specialists, San Dimas, California
  - North American Research Institute, San Dimas, California
  - UCLA, Santa Monica, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Creekside Endocrine Associates, Denver, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - AGA Clinical Trials, Hialeah, Florida
  - Leon Medical Research Corp., Miami, Florida
  - Elite Clinical Research, Miami, Florida
  - DL Research Solutions, Miami, Florida
  - Premier Research Associates, Inc., Miami, Florida
  - Sweet Hope Research Speciality, Inc., Miami Lakes, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Atlanta Center for Clinical Research Nephrology, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - East Coast Institute for Clinical Research, Macon, Georgia
  - East Coast Institute for Research, Macon, Georgia
  - Saltzer Medical Group, Nampa, Idaho
  - Research by Design, LLC, Chicago, Illinois
  - American Health Network of Indiana, Franklin, Indiana
  - My Kidney Center, Manhattan, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Joslin Diabetes Center, Boston, Massachusetts
  - Aa Mrc, Llc, Flint, Michigan
  - St. Louis Heart & Vascular, P.C., St Louis, Missouri
  - NJ Heart, P.A., Linden, New Jersey
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Physicians East Endocrinology, Greenville, North Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - South Carolina Nephrology & Hypertension Center, Orangeburg, South Carolina
  - University of Tennessee Health Science Center at Memphis University Hospital, Memphis, Tennessee
  - Pioneer Research Solutions, Beaumont, Texas
  - Academy of Diabetes, Thyroid and Endocrine, P.A., El Paso, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - Rockwood Medical Center, Fort Worth, Texas
  - Endocrine IPS, PLLC, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - FMC Science, LLC, Lampasas, Texas
  - Clinical Advancement Center PLLC, San Antonio, Texas
  - Briggs Clinical Research, San Antonio, Texas
  - Burke Internal Medicine and Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Northside Endocrinology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanrahan JP, de Boer IH, Bakris GL, Wilson PJ, Wakefield JD, Seferovic JP, Chickering JG, Chien YT, Carlson K, Cressman MD, Currie MG, Milne GT, Profy AT. Effects of the Soluble Guanylate Cyclase Stimulator Praliciguat in Diabetic Kidney Disease: A Randomized Placebo-Controlled Clinical Trial. Clin J Am Soc Nephrol. 2020 Dec 31;16(1):59-69. doi: 10.2215/CJN.08410520. Epub 2020 Dec 16. PMID 33328269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the safety and efficacy of praliciguat (IW-1973) in participants with type 2 diabetes mellitus with albuminuria who were on a stable regimen of renin-angiotensin system inhibitors.
Pre-assignment Details: A total of 156 participants were enrolled in the study.
Groups:
- Placebo: Participants were randomized to receive matching placebo orally for 12 weeks: 1 week of twice daily (BID) dosing (Days 1 through 7) followed by 11 weeks of once daily (QD) dosing.
- Praliciguat 20 mg: Participants were randomized to receive praliciguat 20 milligrams (mg) orally for 12 weeks: 1 week of BID dosing (Days 1 through 7) followed by 11 weeks of QD dosing.
- Praliciguat 40 mg: Participants were randomized to receive praliciguat 40 mg orally for 12 weeks: 1 week of BID dosing (Days 1 through 7) followed by 11 weeks of QD dosing.
Period: Overall Study
Arm/Group | Placebo | Praliciguat 20 mg | Praliciguat 40 mg
Started | 54 | 50 | 52
Completed | 51 | 47 | 42
Not Completed | 3 | 3 | 10
Not completed — Adverse Event | 1 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population consisted of all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Praliciguat 20 mg | Praliciguat 40 mg | Total
Number analyzed (Participants) | 54 | 50 | 52 | 156
Age, Customized [Count of Participants; unit: Participants]
  18 - 45 | 0 | 1 | 2 | 3
  >45 - 65 | 26 | 25 | 23 | 74
  >65 | 28 | 24 | 27 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 20 | 53
  Male | 37 | 34 | 32 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 30 | 30 | 85
  Not Hispanic or Latino | 29 | 20 | 22 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 10 | 13 | 14 | 37
  White | 41 | 33 | 37 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Study Drug-Related TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as those AEs that started or worsened in severity after the initiation of study drug administration. Causality relationship to study drug was per Investigator assessment.
Time Frame: Day 1 up to Day 115
Population: Safety Population consisted of all randomized participants who received at least 1 dose of study drug. Participants in this population were summarized according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Praliciguat 20 mg | Praliciguat 40 mg
Number analyzed (Participants) | 54 | 50 | 52
Participants
  Any TEAE | 24 | 21 | 22
  Study drug-related TEAEs | 6 | 3 | 10

2. Primary Outcome: Percent Change From Baseline in Urine Albumin Creatinine Ratio (UACR) Over Weeks 8 and 12
Description: Urine samples were collected for the analysis of UACR. UACR (milligrams per gram [mg/g]) was calculated as urine albumin (mg per deciliter [mg/dL]) / urine creatinine (g/dL). Change from Baseline was calculated as the average of the UCAR values at Weeks 8 and 12 minus the Baseline value. Data were analyzed using a mixed-effects model repeated measures (MMRM) analysis with change from Baseline in log-transformed UACR as the response variable, treatment, visit, treatment-by visit interaction, and Baseline estimated glomerular filtration rate stratum as fixed effects, Baseline log-transformed UACR and Baseline mean arterial pressure as covariates, and unstructured as the variance-covariance structure.
Time Frame: Baseline; Week 8 to Week 12
Population: Intent-to-Treat Population consisted of all randomized participants who received at least 1 dose of study drug. Participants in this population were evaluated according to the treatment group they were assigned to at Randomization.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Percent Change
Groups:
- Praliciguat Overall: Participants were randomized to receive both 20 mg and 40 mg praliciguat orally for 12 weeks.
Arm/Group | Placebo | Praliciguat 20 mg | Praliciguat 40 mg | Praliciguat Overall
Number analyzed (Participants) | 54 | 50 | 52 | 102
Percent Change | -14.8 [-27.7 to 0.4] | -28.4 [-39.4 to -15.3] | -27.3 [-39.2 to -13.1] | -27.8 [-36.3 to -18.3]
Statistical Analysis 1: Comparison: Placebo vs Praliciguat 20 mg; Treatment comparison between placebo and praliciguat 20 mg. Geometric mean change (%) and the associated confidence intervals (CIs) were derived as 100×[exp(Least Squares Mean Change)-1]; Test type: Superiority; p = 0.2142, Mixed Models Analysis; Geometric mean change (%) = -16.0, 90% CI 2-sided [-33.3 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs Praliciguat 40 mg; Treatment comparison between placebo and praliciguat 40 mg. Geometric mean change (%) and the associated CIs were derived as 100×[exp(Least Squares Mean Change)-1]; Test type: Superiority; p = 0.2718, Mixed Models Analysis; Geometric mean change (%) = -14.6, 90% CI 2-sided [-32.7 to 8.3]
Statistical Analysis 3: Comparison: Placebo vs Praliciguat Overall; Treatment comparison between placebo and praliciguat overall. Geometric mean change (%) and the associated CIs were derived as 100×[exp(Least Squares Mean Change)-1]; Test type: Superiority; p = 0.1736, Mixed Models Analysis; Geometric mean change (%) = -15.3, 90% CI 2-sided [-30.7 to 3.6]

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to Follow-up Visit (Day 115)
Description: TEAEs, defined as those AEs that started or worsened in severity after the initiation of study drug administration are reported for the Safety Population which consisted of all randomized participants who took at least 1 dose of study drug.
Arm/Group | Placebo | Praliciguat 20 mg | Praliciguat 40 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/50 | 4/52
Other Adverse Events (participants affected / at risk) | 24/54 | 21/50 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Praliciguat 20 mg (N=50) | Praliciguat 40 mg (N=52)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Praliciguat 20 mg (N=50) | Praliciguat 40 mg (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03217591/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03217591/SAP_001.pdf